CLINICAL TRIAL: NCT00124254
Title: An Outcome Study of Rheumatoid Hand Arthroplasty
Brief Title: Study of People With Rheumatoid Arthritis Who Require Joint Surgery in the Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Dr. Kevin C. Chung, Professor of Surgery, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR047328 (NIH); R01AR047328 (NIH); 1R01AR047328-01A2 (NIH)
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Arthritis, Rheumatoid
Keywords: Metacarpophalangeal Joint; Arthroplasty; Outcomes; Michigan Hand Outcomes Questionnaire; Joint Replacement
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Surgical group undergoing SMPA
  Interventions: Procedure: Silicone metacarpophalangeal joint arthroplasty
- 2 (Active Comparator): Nosurgical group
  Interventions: Other: Usual care

INTERVENTIONS:
Procedure: Silicone metacarpophalangeal joint arthroplasty — Intervention involves reconstructing the metacarpophalangeal joint using the Swanson silastic implant.
  Other Names: Swanson silastic implant
  Arms: 1
Other: Usual care — Non-surgical usual care
  Arms: 2

SUMMARY:
A procedure called silicone metacarpophalangeal joint arthroplasty (SMPA) is sometimes used to treat knuckle deformity in the hands of rheumatoid arthritis (RA) patients. The purpose of this study is to compare the health outcomes of RA patients who choose to undergo SMPA surgery to RA patients who do not undergo surgery.

DETAILED DESCRIPTION:
The purpose of this study is to provide a better understanding of the effectiveness of SMPA, a procedure to correct knuckle deformity in the hands of rheumatoid arthritis patients. This study will examine whether rheumatoid arthritis patients who undergo SMPA will have better outcomes than those patients who do not have this surgery.

RA affects 2.1 million Americans and costs the United States an estimated $8.7 billion annually in medical costs and wages. RA is a progressive disease, and approximately 25% of RA patients experience hand deformities associated with the destruction of the metacarpophalangeal (MCP) joints. For the past 30 years, SMPA has been performed on such patients to correct metacarpophalangeal joint deformity in the rheumatoid hand. SMPA can provide pain relief, restoration of function, and aesthetic improvement to the patient. However, because data are limited on its efficacy, SMPA remains a controversial procedure. Hand surgeons and rheumatologists frequently disagree about the indications for this procedure and its value to their patients. In addition, most published studies have been hampered by inadequate consideration of research design, small sample size, and inconsistent outcome measures. The purpose of this study is to measure short- and long-term outcomes following SMPA. The study will also define indications of the surgery for specific patient groups and disease severity. The experiences of both surgery and rheumatology services will be used to jointly evaluate this surgical procedure.

This study is a multicenter, international outcomes study to evaluate RA patients with severe MCP joint problems. Patients will choose to be enrolled into a surgical group undergoing SMPA or a nonsurgical group. Patients will be evaluated at Month 6 and annually until the third year. Patient evaluations will be based on the Michigan Hand Outcomes Questionnaire, the Arthritis Impact Measurement Scales questionnaire, and standard, objective hand function tests.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis based on the diagnostic criteria of the American Rheumatology Association
* Able to complete questionnaires in English
* Sum of average metacarpophalangeal joint ulnar drift AND average metacarpophalangeal joint extensor lag of 50 degrees or greater

Exclusion Criteria:

* Severe medical condition precluding surgery
* Concomitant extensor tendon ruptures and metacarpophalangeal joint disease
* Other joint injury of the hand (e.g., swan-neck deformity, boutonniere deformity) requiring surgery
* Previous metacarpophalangeal joint replacement on their study hand
* Disease modifying antirheumatic drugs (DMARDs) within the 3 months prior to study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2003-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Michigan Hand Outcomes Questionnaire | Baseline, 6 months, 1 year, 2 years, 3 year

SECONDARY OUTCOMES:
Arthritis Impact Measurement Scales Questionnaire | Baseline, 6 months, 1 year, 2 years, 3 years
Standard, objective hand function tests | Baseline, 6 months, 1 year, 2 years, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C. Chung, MD, MS, Principal Investigator — University of Michigan
Locations (3):
- United States (2):
  - Curtis National Hand Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
- Pulvertaft Hand Centre, Derby, United Kingdom

REFERENCES:
- [Background] Mathews AL, Burns PB, Chung KC. How Rheumatoid Arthritis Patients Make Decisions Regarding Hand Reconstruction: A Qualitative Study from the Silicone Arthroplasty in Rheumatoid Arthritis Project. Plast Reconstr Surg. 2016 May;137(5):1507-1514. doi: 10.1097/PRS.0000000000002083. PMID 26796370
- [Background] Sears ED, Burns PB, Chung KC. Relationship between Patient Expectations and Clinical Measures in Patients Undergoing Rheumatoid Hand Surgery from the Silicone Arthroplasty in Rheumatoid Arthritis (SARA) Study. Plast Reconstr Surg. 2015 Dec;136(6):775e-781e. doi: 10.1097/PRS.0000000000001778. PMID 26595031
- [Background] Mathews AL, Coleska A, Burns PB, Chung KC. Evolution of Patient Decision-Making Regarding Medical Treatment of Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2016 Mar;68(3):318-24. doi: 10.1002/acr.22688. PMID 26315611
- [Background] Squitieri L, Chung KC, Hutton DW, Burns PB, Kim HM, Mahmoudi E. A 5-Year Cost-Effectiveness Analysis of Silicone Metacarpophalangeal Arthroplasty in Patients with Rheumatoid Arthritis. Plast Reconstr Surg. 2015 Aug;136(2):305-314. doi: 10.1097/PRS.0000000000001409. PMID 25909303
- [Background] Chung KC, Nellans KW, Burns PB, Wilgis EF, Burke FD, Fox DA, Kim HM. Patient expectations and long-term outcomes in rheumatoid arthritis patients: results from the SARA (Silicone Arthroplasty in Rheumatoid Arthritis) study. Clin Rheumatol. 2015 Apr;34(4):641-51. doi: 10.1007/s10067-014-2775-z. Epub 2014 Sep 30. PMID 25267562
- [Background] Chetta M, Burns PB, Kim HM, Burke FD, Wilgis EFS, Fox DA, Chung KC. The effect of swan neck and boutonniere deformities on the outcome of silicone metacarpophalangeal joint arthroplasty in rheumatoid arthritis. Plast Reconstr Surg. 2013 Sep;132(3):597-603. doi: 10.1097/PRS.0b013e31829ad1c1. PMID 23985634
- [Background] Chung KC, Burns PB, Kim HM, Burke FD, Wilgis EF, Fox DA. Long-term followup for rheumatoid arthritis patients in a multicenter outcomes study of silicone metacarpophalangeal joint arthroplasty. Arthritis Care Res (Hoboken). 2012 Sep;64(9):1292-300. doi: 10.1002/acr.21705. PMID 22511483
- [Background] Chung KC, Burns PB, Reichert HA, Fox DA, Burke FD, Wilgis EF, Regan M, Kim HM. Properties of the International Classification for Functioning, Disability and Health in assessing hand outcomes in patients with rheumatoid arthritis. J Rehabil Med. 2011 Mar;43(4):292-8. doi: 10.2340/16501977-0671. PMID 21267527
- [Background] Waljee JF, Chung KC, Kim HM, Burns PB, Burke FD, Wilgis EF, Fox DA. Validity and responsiveness of the Michigan Hand Questionnaire in patients with rheumatoid arthritis: a multicenter, international study. Arthritis Care Res (Hoboken). 2010 Nov;62(11):1569-77. doi: 10.1002/acr.20274. Epub 2010 Jun 2. PMID 20521331
- [Background] Chung KC, Kotsis SV, Fox DA, Regan M, Burke FD, Wilgis EF, Kim HM. Differences between the United States and the United Kingdom in the treatment of rheumatoid arthritis: analyses from a hand arthroplasty trial. Clin Rheumatol. 2010 Apr;29(4):363-7. doi: 10.1007/s10067-009-1314-9. PMID 20077124
- [Background] Chung KC, Kotsis SV, Wilgis EF, Fox DA, Regan M, Kim HM, Burke FD. Outcomes of silicone arthroplasty for rheumatoid metacarpophalangeal joints stratified by fingers. J Hand Surg Am. 2009 Nov;34(9):1647-52. doi: 10.1016/j.jhsa.2009.06.029. PMID 19896008
- [Background] Chung KC, Burke FD, Wilgis EFS, Regan M, Kim HM, Fox DA. A prospective study comparing outcomes after reconstruction in rheumatoid arthritis patients with severe ulnar drift deformities. Plast Reconstr Surg. 2009 Jun;123(6):1769-1777. doi: 10.1097/PRS.0b013e3181a65b5a. PMID 19483578
- [Result] Chung KC, Kotsis SV, Kim HM. A prospective outcomes study of Swanson metacarpophalangeal joint arthroplasty for the rheumatoid hand. J Hand Surg Am. 2004 Jul;29(4):646-53. doi: 10.1016/j.jhsa.2004.03.004. PMID 15249089
- [Result] Chung KC, Kotsis SV, Kim HM, Burke FD, Wilgis EF. Reasons why rheumatoid arthritis patients seek surgical treatment for hand deformities. J Hand Surg Am. 2006 Feb;31(2):289-94. doi: 10.1016/j.jhsa.2005.10.005. PMID 16473693
- [Result] Mandl LA, Burke FD, Shaw Wilgis EF, Lyman S, Katz JN, Chung KC. Could preoperative preferences and expectations influence surgical decision making? Rheumatoid arthritis patients contemplating metacarpophalangeal joint arthroplasty. Plast Reconstr Surg. 2008 Jan;121(1):175-180. doi: 10.1097/01.prs.0000295376.70930.7e. PMID 18176218